CLINICAL TRIAL: NCT03945812
Title: The Impact of Using Platelet-Rich Plasma Versus Granulocyte Colony-Stimulating Factor Versus Placebo on the Outcomes of Frozen Embryo Transfer: A Double Blind Randomized Controlled Trial
Brief Title: Platelet-Rich Plasma vs. Granulocyte Colony-Stimulating Factor vs. Placebo and Outcomes in Frozen Embryo Transfer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wael Elbanna Clinic (Other)
Collaborators: National Research Centre, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INDV-0909012
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Infertility; Frozen Embryo Transfer (FET)
Keywords: GCSF; PRP; Pregnancy
MeSH Terms: conditions — Infertility | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Granulocyte Colony Stimulating Factor Arm (Active Comparator): Women in this group will receive GCSF with conventional hormonal therapy:
  Estradiol valerate 6mg/day from day 2 of menstrual cycle Vaginal sildenafil citrate 25mg / 6 hours Then frozen embryo transfer will be performed.
  Interventions: Drug: Granulocyte Colony Stimulating Factor
- Platelet Rich Plasma Arm (Active Comparator): Women in this group will receive PRP with conventional hormonal therapy:
  Estradiol valerate 6mg/day from day 2 of menstrual cycle Vaginal sildenafil citrate 25mg / 6 hours Then frozen embryo transfer will be performed.
  Interventions: Other: Platelet Rich Plasma Arm
- Saline (Placebo Comparator): Women in this group will receive saline with conventional hormonal therapy:
  Estradiol valerate 6mg/day from day 2 of menstrual cycle Vaginal sildenafil citrate 25mg / 6 hours Then frozen embryo transfer will be performed.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Granulocyte Colony Stimulating Factor — Filgrastim, Amgen, California, USA 300 mg/1.0 mL
  Other Names: Filgrastim
  Arms: Granulocyte Colony Stimulating Factor Arm
Other: Platelet Rich Plasma Arm — Platelet Rich Plasma Arm
  Arms: Platelet Rich Plasma Arm
Other: Saline — Saline 9%
  Other Names: Saline 9%
  Arms: Saline

SUMMARY:
The goal of this clinical trial is to assess the impact of using Platelet-Rich Plasma (PRP) vs. Granulocyte Colony-Stimulating Factor (GCSF) vs. placebo on the outcomes of frozen embryo transfer (FET) in terms of clinical pregnancy rates. It will also assess their effect on chemical pregnancy rate, implantation rate, delivery outcomes, and endometrial parameters.

The main questions it aims to answer are:

Do the clinical pregnancy rates differ upon using PRP vs. GCSF vs. placebo during FET? What are the effects of PRP vs. GCSF vs. placebo during FET on chemical pregnancy rate, implantation rate, delivery outcomes, and endometrial parameters?

Researchers will compare the effect of administration of PRP vs. GCSF vs. placebo during FET on pregnancy outcomes.

Participants will be randomized to receive the study intervention seven days before embryo transfer: 1.0 ml of either PRP (prepared in-house), GCSF (Filgrastim, 300 mcg/1.0 mL), or 0.9% saline (placebo). The intervention will be administered by slow infusion into the uterine cavity with an intrauterine insemination catheter.

DETAILED DESCRIPTION:
INTRODUCTION AND STUDY RATIONALE Despite the advancements in the treatment of infertility, repeated failure of implantation continues as a challenging difficulty.

Embryo implantation is affected by many factors. Many efforts were made to improve the implantation rate by different methods blastocyst transfer, assisted hatching, preimplantation genetic screening, hysteroscopy, removal of hydrosalpinges and endometrial scratch. Furthermore, infertility specialists suggested some empirical methods like the infusion in the uterine cavity of platelet-rich plasma (PRP) in patients with thin endometrium which has been shown to be effective in improving the pregnancy rate.

Another factor is granulocyte colony stimulating factor (GCSF) which has receptors in endometrial cells and may have a role in implantation. The use of GCSF in assisted reproductive technology (ART) has been tried by many research studies either via intrauterine or systemic administration.

There are limited studies that compared the impact of PRP and GCSF administration on the pregnancy rate and on the endometrial thickness with a small sample size.

The rationale behind this current study is to assess the impact of using PRP versus GCSF versus on the outcomes of FET in terms of pregnancy rates.

STUDY OBJECTIVES

Primary:

The primary objective of the study is to compare the clinical pregnancy rate determined by presence of fetal heart beat in transvaginal ultrasound after 6 weeks of embryo transfer in all groups.

Secondary:

To compare the following in the three study arms:

* Chemical pregnancy determined by positive serum β-HCG, 2 weeks after embryo transfer.
* Delivery outcomes: miscarriage and live bith rates.
* The implantation rate, calculated by dividing the number of gestational sacs observed via ultrasound by the number of embryos transferred.
* The change in endometrial parameters, assessed as endometrial thickness, Doppler indices, endometrial vascularization, blood volume histogram indices, and the histological dating of the endometrium.

SAMPLE SIZE CALCULATION The sample size was calculated using G*Power 3.1.9.7. Based on Jie Li et al. study, the clinical pregnancy rate in the GCSF group was 25.1% compared to 14.4% in the placebo or no-treatment group. Assuming a 10% improvement in the clinical pregnancy rate with GCSF, a two-sided alpha level of 5%, and achieving 80% power, the sample size was initially calculated to be 498 women. To account for a 25% anticipated dropout rate, the final sample size was adjusted to 624 women (208 in each group). Although no studies comparing PRP to placebo, specifically in our study population, were published before designing our study, a 22% improvement in the clinical pregnancy rate with PRP was observed in studies involving women with thin endometrium. To reach sufficient power to detect differences between the three study arms, our calculation was based on GCSF.

Li J, Mo S, Chen Y. The effect of G-CSF on infertile women undergoing IVF treatment: A meta-analysis. Systems Biology in Reproductive Medicine. 2017/07/04 2017;63(4):239-247. doi:10.1080/19396368.2017.1287225

STATISTICAL ANALYSIS We will compare participants' baseline demographics and clinical characteristics across the study's three arms: PRP, GCSF, and saline. Categorical variables will be presented as frequency and percentage and compared using the Chi-squared test (χ2). Normally distributed variables will be reported as mean (standard deviation; SD) and compared using one-way analysis of variance (ANOVA), while non-normally distributed will be reported as median (25th to 75th percentile) and compared using the Kruskal-Wallis test. A p-value of less than 0.05 will be considered statistically significant.

Clinical pregnancy rate will be adjusted by the endometrial thickness (thin versus normal (≥ 7 mm)) in all groups.

An interim analysis will be conducted by the Data Monitoring Committee (DMC) after 60% of participants have been enrolled in the study to assess the efficacy of the intervention arms.

SUB-GROUP ANALYSIS: to evaluate the clinical pregnancy rates among patients based on:

* Anti-Müllerian hormone (AMH) value <1 ng/ml (poor responders)
* Preimplantation genetic screening (PGS)
* Reepeated, two or more, failed implantations (RIF).
* Triple-layered endometrium, evaluated by TVUS in the mid-luteal phase.

ELIGIBILITY:
Inclusion Criteria:

* All women aged 20-40 years
* Non-smoker
* BMI < 30
* Normal endometrial cavity confirmed by hysteroscopy and ultrasound
* Visiting the center for IVF by FET during the period of the study

Exclusion Criteria:

* History of anti-phospholipid syndrome confirmed by serological tests.
* History of any hematological and immunological disorders
* History of chromosomal or genetic abnormalities in the patient or in the family
* Any uterine abnormalities (congenital or acquired)
* Previous uterine surgeries except caesarean section
* Hypersensitivity to G-CSF
* Uncontrolled systemic disease

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 665 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
The clinical pregnancy rate | 6 to 8 weeks of embryo transfer
  Definition: The presence of fetal heartbeats in transvaginal ultrasound after 6 to 8 weeks of embryo transfer in all groups.
  Unit of Measure: The percentage of participants who will achieve a clinical pregnancy among those who underwent the embryo transfer, calculated by dividing the number of participants who will have a clinical pregnancy by the total number of participants who underwent embryo transfer and multiplying by 100.

SECONDARY OUTCOMES:
Chemical pregnancy rate | 2 weeks post embryo transfer
  Definition: Positive serum β-hCG 2 weeks post-embryo transfer.
  Unit of Measure: The percentage of participants who will achieve a chemical pregnancy among those who underwent the embryo transfer, calculated by dividing the number of participants who will have a chemical pregnancy by the total number of participants who underwent embryo transfer and multiplying by 100.
Miscarriage rate | 20 weeks of gestation
  Definition: Loss of a clinical pregnancy before 20 weeks of gestation.
  Unit of Measure: The percentage of participants who will have a miscarriage among those who achieved clinical pregnancy, calculated by dividing the number of participants who will have a miscarriage by the total number of participants who achieved clinical pregnancy and multiplying by 100.
Live-birth rate | The live birth rate is assessed at the time of birth, including both full-term and preterm live births.
  Definition: the number of deliveries that resulted in a live-born neonate.
  Unit of Measure: The percentage of participants who will have a live-born neonate among those who achieved clinical pregnancy, calculated by dividing the number of participants who will have a live-born neonate by the total number of participants who achieved clinical pregnancy and multiplying by 100.
Implantation rate | Between 3 and 5 weeks after embryo transfer.
  Definition: Number of gestational sacs observed via transvaginal ultrasound divided by number of embryos transferred.
  Unit of Measure: Ratio (sacs/embryos)
Endometrial Thickness | The changes in endometrial parameters between the intervention cycle and the natural cycle will be measured during the mid-luteal phase (during 18-23 days of the cycle).
  Endometrial thickness is measured as the maximum anterior-posterior thickness (in mm) of the endometrial echo on a long-axis transvaginal view of the uterus using transvaginal ultrasound.
Uterine Artery Doppler Indices (e.g., PI, RI) | The changes in endometrial parameters between the intervention cycle and the natural cycle will be measured during the mid-luteal phase (during 18-23 days of the cycle).
  Assessment of uterine artery blood flow resistance using Doppler ultrasound. Pulsatility Index (PI) and Resistance Index (RI) are the main Doppler indices used. Units: Both PI and RI are dimensionless (no units), as they are ratios derived from velocity measurements. Typical reporting: PI and RI are given as numeric values (e.g., PI = 1.75, RI = 0.72).
Endometrial Vascularization | The changes in endometrial parameters between the intervention cycle and the natural cycle will be measured during the mid-luteal phase (during 18-23 days of the cycle).
  Endometrial Vascularization Tool: 3D Power Doppler histogram. Measured as: Microvessel Density (MVD) and Vascular Endothelial Growth Factor (VEGF) expression. Units: MVD; number of microvessels per square millimeter, VEGF H-score; semi-quantitative, unitless score based on staining intensity.
  Blood Volume Histogram Indices: Vascularization Index (VI), Flow Index (FI), Vascularization-Flow Index (VFI) are the main indices. Units: These indices are dimensionless (unitless ratios or percentages) as they are calculated from the proportion or intensity of power Doppler signals within a defined volume.
Histogram Indices (Blood flow velocities) | The changes in endometrial parameters between the intervention cycle and the natural cycle will be measured during the mid-luteal phase (during 18-23 days of the cycle).
  Definition: Histograms in medical imaging often display the distribution of blood flow velocities.
  Units: cm/s or mL/min (velocity or volume flow rate).
Histogram Indices (cell sizes) | The changes in endometrial parameters between the intervention cycle and the natural cycle will be measured during the mid-luteal phase (during 18-23 days of the cycle).
  Definition: Histograms in medical imaging often display the distribution of cell sizes.
  Units: femtoliters (fL) for mean cell volume
Histological Dating of Endometrium | The changes in endometrial parameters between the intervention cycle and the natural cycle will be measured during the mid-luteal phase (during 18-23 days of the cycle).
  Microscopic assessment to determine phase consistency with expected luteal day using histological biopsy, assessed via Noyes criteria. Unit: Luteal phase date match (yes/no or deviation in days). Units: Days of the menstrual cycle (e.g., Day 17, Day 19), or described by phase (proliferative, secretory, etc.). No physical units are assigned to histological dating; it is a temporal or qualitative assessment based on morphological criteria

CONTACTS AND LOCATIONS:
Overall Officials: Wael SS Elbanna, Consultant, Principal Investigator — Wael Elbanna Clinic
Locations (1):
- Hayat center, Maadi, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehrafza M, Kabodmehri R, Nikpouri Z, Pourseify G, Raoufi A, Eftekhari A, Samadnia S, Hosseini A. Comparing the Impact of Autologous Platelet-rich Plasma and Granulocyte Colony Stimulating Factor on Pregnancy Outcome in Patients with Repeated Implantation Failure. J Reprod Infertil. 2019 Jan-Mar;20(1):35-41. PMID 30859080
- [Background] Coughlan C, Ledger W, Wang Q, Liu F, Demirol A, Gurgan T, Cutting R, Ong K, Sallam H, Li TC. Recurrent implantation failure: definition and management. Reprod Biomed Online. 2014 Jan;28(1):14-38. doi: 10.1016/j.rbmo.2013.08.011. Epub 2013 Sep 14. PMID 24269084
- [Background] Rinehart J. Recurrent implantation failure: definition. J Assist Reprod Genet. 2007 Jul;24(7):284-7. doi: 10.1007/s10815-007-9147-4. Epub 2007 Aug 3. PMID 17674185
- [Background] Chang Y, Li J, Chen Y, Wei L, Yang X, Shi Y, Liang X. Autologous platelet-rich plasma promotes endometrial growth and improves pregnancy outcome during in vitro fertilization. Int J Clin Exp Med. 2015 Jan 15;8(1):1286-90. eCollection 2015. PMID 25785127